CLINICAL TRIAL: NCT06564194
Title: A Phase 1 Randomized, Double-Blinded Study to Assess the Safety, Reactogenicity and Immunogenicity of JCXH-108, an mRNA-based Investigational Vaccine Against Respiratory Syncytial Virus (RSV) in Healthy Subjects ≥ 60 Years of Age and 18-45 Years of Age
Brief Title: A Phase 1 Study to Evaluate JCXH-108, an mRNA-based Vaccine Against RSV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immorna Biotherapeutics, Inc. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JCXH-108-001
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Syncytial Virus (RSV); Infectious Disease
Keywords: mRNA vaccine; RSV vaccination; Healthy subjects
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational product (Experimental): Subjects randomized to this arm will be given the investigational product (JCXH-108).
  Interventions: Biological: JCXH-108
- Placebo (Placebo Comparator): Subjects randomized to this arm will be given a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: JCXH-108 — IM injection
  Arms: Investigational product
Other: Placebo — IM injection
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the safety, reactogenicity and immunogenicity of an mRNA-based vaccine, JCXH-108, the prevention of Respiratory Syncytial Virus (RSV) infection and diseases.

Participants will be randomized to receive either JCXH-108 or placebo.

DETAILED DESCRIPTION:
This Phase 1 study plans to enroll a total of 75 participants.

Three cohorts with two different dose levels will be explored and each cohort will enroll 25 participants. Participants in each cohort will be randomized (4:1) to receive either JCXH-108 (n=20) or placebo (normal saline, n=5). A low dose of JCXH-108 will be explored vs placebo in the 18-45 years of age group first. A high dose will be explored vs placebo in the 18-45 years and ≥ 60 years of age groups once safety data is reviewed for the Sentinel subjects in the low dose cohort. The dose level of JCXH-108 will depend on the time the participant joins the study. Each participant will receive a single dose of JCXH-108 administered intramuscularly (IM) on day 1.

ELIGIBILITY:
Main Inclusion Criteria:

* Sex: Male or female; female subjects may be of childbearing potential or postmenopausal.
* Age: 18-45 years of age or ≥ 60 years of age at screening
* Status: Healthy subjects.
* Subjects must agree to not be vaccinated with any RSV vaccine while participating in this study.
* Subjects must agree to not be vaccinated with any RNA-based vaccines 30 days before D1 through 30 days after D1.

Main Exclusion Criteria:

* Subjects with current diagnosis of RSV infection or diseases.
* Previous vaccination against RSV.
* Subjects with any respiratory illness deemed clinically relevant by the Investigator within the past month OR hospitalization >24 hours for any reason within the past month prior to Day 1.
* Subjects with history of myocarditis or pericarditis, or with adverse events (AEs) after mRNA vaccination that are in nature and severity beyond the common expected AEs necessitating medical intervention.
* Subjects who received any non-live vaccine within 14 days prior to Day 1.
* Subjects who received within 28 days prior to Day 1: (1) Any live vaccine, (2) Immunomodulators or immune-suppressive medication, (3) Granulocyte or granulocyte-macrophage colony-stimulating factor, and (4) Three or more consecutive days of systemic corticosteroids. Note: subjects on stable dose of steroid replacement (for chronic disease such as iatrogenic deficiency) of prednisone ≤10 mg/day or equivalent are allowed.
* Subjects who currently receive other investigational agents or devices.
* Subjects with active or suspected immunosuppression, immunodeficiency, asplenia, recurrent severe infections or autoimmune diseases. Certain immune-mediated conditions (e.g., Hashimoto thyroiditis) that are well controlled and stable are allowed.
* Subjects receiving systemic antiviral therapy.
* Subjects with a positive screening test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or anti-human HIV-1 and 2 antibodies, syphilis.
* Subjects with a positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening or on Day 1 prior to vaccine administration (JCXH-108 or placebo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
SAE Frequency | Day 1 - Day 180 (6 Months)
  Frequency of SAEs characterized by type, severity, duration, and relationship to the JCXH-108 recorded from Day 1 (D1) post-vaccine administration through follow-up completion.
Injection site reaction | Day 1 - Day 30
  Solicited local injection site reactions characterized by frequency, severity, and duration recorded within 30 days after administration after vaccine administration (JCXH-108 or Placebo)
Solicited systemic reaction frequency | Day 1 - Day 30
  Solicited systemic adverse reactions characterized by frequency, severity, and duration recorded within 30 days after vaccine administration (JCXH-108 or Placebo)
AE frequency | Day 1 -Day 30
  Adverse events (AEs) including unsolicited AEs characterized by type, severity, duration, and relationship to the vaccine (JCXH-108 or Placebo) recorded from Day 1 post-vaccine administration to within 30 days following vaccine administration
Medically attended AE frequency | Day 1 - Day 180 (6 Months)
  Medically attended AEs (MAAEs) characterized by frequency, severity, duration, and relationship to the vaccine (JCXH-108 or Placebo) recorded from Day 1 post-vaccine administration (JCXH-108 or Placebo) through follow-up completion
Potential immune-mediated adverse events frequency | Day 1 - Day 180 (6 Months)
  Potential immune-mediated disease (pIMDs) characterized by frequency, severity, duration, and relationship to the vaccine (JCXH-108 or Placebo) recorded from Day 1 post-vaccine administration (JCXH-108 or Placebo) through follow-up completion

SECONDARY OUTCOMES:
RSV-A and RSV-B antibody levels | Day 1 - Day 180 (6 Months)
  Levels of serum neutralizing antibodies against RSV-A and RSV-B as compared to Day 1 pre-dose (baseline) at Day 29, Month 3 and Month 6 after the vaccine administration
IgG antibody levels | Day 1 - Day 30
  Levels of serum RSV pre-F antibodies of IgG1, IgG2, IgG3, and IgG4 as compared to Day 1 pre-dose (baseline) at Day 29, after the vaccine administration. Measured in women of childbearing potential only.

OTHER OUTCOMES:
T-cell responses | Day 1 -Day 180 (6 Months)
  T-cell responses to vaccine-encoded antigen in peripheral blood mononuclear cells (PBMCs) determined by enzyme-linked immunosorbent spot (ELISpot) and Intracellular Cytokine Staining (ICS) assays, as compared to baseline (Day 1 pre-dose) at 29 days and 6 months after the vaccine administration (Day 30 and Month 6).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Health Awareness, Jupiter, Florida
  - DelRicht - New Orleans, New Orleans, Louisiana
  - Sundance Clinical Research, St Louis, Missouri